CLINICAL TRIAL: NCT03286582
Title: A Randomized, Open-Label, Controlled Trial of Topical AC-203 in Subjects With Bullous Pemphigoid
Brief Title: A Proof-of-Concept Study of Topical AC-203 in Patients With Bullous Pemphigoid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated with partial enrollment completed
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-203-BP-001
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — diacerein; Ointments; Clobetasol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AC-203 (Experimental)
  Interventions: Drug: AC-203 1% Topical Ointment
- Clobetasol (Active Comparator)
  Interventions: Drug: Clobetasol 0.05% Topical Ointment

INTERVENTIONS:
Drug: AC-203 1% Topical Ointment — AC-203 1% ointment BID (twice daily)
  Arms: AC-203
Drug: Clobetasol 0.05% Topical Ointment — Clobetasol 0.05% Topical Ointment BID
  Arms: Clobetasol

SUMMARY:
Bullous pemphigoid (BP) is a chronic, inflammatory, subepidermal, autoimmune blistering disease which mainly develops in the elderly, with onset usually in the late 70s and a substantial increase in incidence in people older than 80 years. If untreated, it can persist for months or years, with periods of spontaneous remissions and exacerbations. It has been found that blisters and sera of BP patients contain abnormally high levels of pro-inflammatory cytokines such as interleukin-6 (IL-6) and IL-8. Recently, it also has been demonstrated that NLRP3 (NACHT, LRR and PYD domains-containing protein 3) inflammasome components (the NLRP3-caspase-1-IL-18 axis) were significantly up-regulated in peripheral blood mononuclear cells from BP patients and positively correlated with disease activity. AC-203 is a topical formulation of an oral modulator of inflammasome and IL-1beta pathways. In vitro studies have demonstrated that AC-203 significantly reduced secretion of IL-6 and moderately reduced IL-8 secretion in HaCaT cells treated with specific anti-BP180 IgG. This study is designed to test the safety, tolerability, efficacy, and pharmacokinetics of AC-203 ointment (vs. a topical steroid comparator representing standard of care) ointment in subjects with BP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 to 90 years old, inclusive, at enrollment.
2. Diagnosis of bullous pemphigoid confirmed by histopathology and one of following assessments:

   1. Direct immunoﬂuorescence (DIF)
   2. Indirect immunoﬂuorescence (IIF)
   3. ELISA test (ELISA detection of immunoglobulin G (IgG) anti-BP180 autoantibodies in serum more than 9 U/mL).
3. Localized or limited BP with the occurrence of <10 new blisters per day in the week prior to enrollment.
4. Is male, or is female and meets all the following criteria:

   1. Not breastfeeding
   2. If of childbearing potential (defined as non-post hysterectomy or non-post-menopausal [≥50 years of age and amenorrheic for at least 1 year]), must have a negative pregnancy test result (human chorionic gonadotropin, beta subunit [bhCG]) at Visit 1, and must practice and be willing to continue to practice appropriate birth control (abstinence, double barrier methods, hormonal contraceptives, intrauterine device, or tubal ligation) during the entire duration of the study
5. Is able to understand and sign the Informed Consent Form (ICF), communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

1. Diagnosis of pemphigus, dermatitis, eczema, psoriasis, or other skin condition which in the opinion of the investigator may confound diagnosis, treatment, or evaluation of bullous pemphigoid.
2. Use of oral steroids in the 2 weeks prior to enrollment at a dose greater than prednisolone equivalent dose (PED) of 10 mg/day.
3. Use of topical steroids for more than 3 consecutive days in the 2 weeks prior to enrollment.
4. Use of non-steroid immunosuppressants including but not limited to azathioprine, mycophenolate, cyclophosphamide, chlorambucil, methotrexate, tacrolimus, or cyclosporine in the 2 weeks prior to enrollment.
5. Use of systemic antibiotics in the 2 weeks prior to enrollment.
6. Use of oral dapsone in the 2 weeks prior to enrollment.
7. Treatment with intravenous immunoglobulin (IVIG) in the 8 weeks prior to enrollment.
8. Any prior use of approved or investigational biologic anti-inflammatory therapy within 6 months prior to enrollment, including but not limited to: anakinra, rilonacept, canakinumab, etanercept, adalimumab, infliximab, rituximab, certolizumab, golimumab, tocilizumab, bertilimumab, or abatacept.
9. Presence of active systemic infections.
10. Any clinically significant medical condition or laboratory value that could potentially affect study participation and/or personal well-being, as judged by the investigator.
11. History of allergy or hypersensitivity to any component of study medication or clobetasol.
12. Has participated in a clinical study within 30 days prior to enrollment.
13. Is an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the clinical study site, or is directly affiliated with the study at the clinical study site.
14. Is employed by the sponsor (i.e., is an employee, temporary contract worker, or designee responsible for the conduct of the study).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events during the treatment period | 10 Weeks

SECONDARY OUTCOMES:
Proportion achieving disease control (no new blisters within prior week) | 2, 4, 5, 6, 8, 10 Weeks
New blister count | 2, 4, 5, 6, 8, 10 Weeks
Time to disease control | 2, 4, 5, 6, 8, 10 Weeks
Proportion of subjects who require rescue therapy prior to Week 6 | 2, 4, 5, 6 Weeks
BPDAI (BP Disease Area Index) score | 2, 4, 5, 6, 8, 10 Weeks
Pruritus VAS (Visual Analogue Scale) score change from baseline | 2, 4, 5, 6, 8, 10 Weeks
DLQI (Dermatology Life Quality Index) score change from baseline | 6, 10 Weeks
Inflammation marker | 6 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho YT, Lee CH, Lee JY, Chu CY. Targeting antibody-mediated complement-independent mechanism in bullous pemphigoid with diacerein. J Dermatol Sci. 2024 Apr;114(1):44-51. doi: 10.1016/j.jdermsci.2024.03.001. Epub 2024 Mar 6. PMID 38508975